CLINICAL TRIAL: NCT01998269
Title: A Mixed Methods Approach to the Development and Testing of the Measure of Drug Self-Management (MeDS), an Assessment for Use in Clinical Settings Among English and Spanish-speaking Patients With Hypertension and Diabetes.
Brief Title: A Mixed Methods Approach to the Development and Testing of the Measure of Drug Self-Management (MeDS)
Acronym: MeDS
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3049
Record Dates: First submitted 2013-11-15; First posted 2013-11-28 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients with diabetes and hypertension

SUMMARY:
The study objective is to develop and test a Measure of Drug Self-Management for use in clinical settings among patients with hypertension and diabetes.

While medication non-adherence is a highly recognized public health and patient safety concern, it is rarely assessed in a routine and consistent manner in clinical settings. With the aging of the US population and rising rates of chronic disease, an increasing number of adults are being prescribed multi-drug regimens that require greater self-management skills. Despite the complexity of medication use, adherence has most commonly been measured as a limited set of behaviors (i.e., filling a prescription, taking doses). This emphasis has, over time, simplified how we think of prescription (Rx) medication use and directed attention away from the full range of tasks associated with effective Rx self-management. The field of health literacy research has deconstructed these tasks in considerable detail in recent years, and can offer insight into a more comprehensive measurement of patients' outpatient Rx use.

There is a clear need for a brief, yet inclusive, measure of adherence that can be used in clinical settings to routinely assess patients' use of complex Rx regimens. Such an assessment could be used to guide clinicians in addressing specific patient challenges to safe and appropriate medication use. In response to this need, our study proposes to develop a new assessment of medication self-management. This unique measure will utilize health literacy best practices to promote patient comprehension and ease-of-use; it will also be tailored to patients' actual regimens via electronic health record (EHR) data. Finally, the tool will be available in both English and Spanish to support use among diverse patient populations. Our study aims are to:

1. Develop and refine a Measure of Drug Self-Management (MeDS) prototype.
2. Inform the content, structure and delivery of the MeDS through targeted discussions with patients, providers and information technology specialists.
3. Test the reliability and validity of the MeDS among patients with diabetes and hypertension

H1: The MeDS will strongly correlate with other self-report adherence measures.

ELIGIBILITY:
Inclusion Criteria:

* be ≥ 18 years old,
* have a diagnosis of diabetes and hypertension,
* be prescribed 3 or more drugs to treat these conditions,
* speak English or Spanish as their primary language,
* have primary responsibility for administering their own medications,
* be a registered UNC patient.

Exclusion Criteria:

* severe, uncorrectable visual, hearing or cognitive impairments that would preclude study consent or participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, primary care patients with diabetes and hypertension
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy C Bailey, PhD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Ambulatory Care Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 210 patients were recruited from the University of North Carolina Ambulatory Care Center. 17 patients participated in focus groups to help develop the medication self-management tool (MeDS tool). The other 193 participated in item performance testing. The results of item performance testing are reported here.
Groups:
- Adult Patients With Diabetes and Hypertension: English-speaking, adult patients with diabetes and hypertension. There are no study arms - this was a cross-sectional study to develop and validate a measure of medication self-management skills. A total of 210 patients were recruited. 17 participated in focus groups to help develop the tool. The other 193 participated in item performance testing. The results of item performance testing are reported here.
Period: Overall Study
Arm/Group | Adult Patients With Diabetes and Hypertension
Started | 193
Completed | 193
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adult Patients With Diabetes and Hypertension: There are no study arms. This was a cross-sectional study to develop a scale.
Arm/Group | Adult Patients With Diabetes and Hypertension
Number analyzed (Participants) | 193
Age, Continuous [Mean (Full Range); unit: years] | 61.1 [28 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 105
  White | 83
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Measure of Medication Self-Management (MeDS)
Description: The MeDS is an assessment of medication self-management skills. The MeDS tool has 14 questions, the minimum score is 0 (poor medication self-management skills) and the maximum score is 14 (adequate self-management skills). The internal consistency of the scale is .72 (cronbach's alpha), which is considered adequate internal consistency. The MeDS was compared to The Morisky Medication Adherence Scale is one of the most commonly used assessments of medication adherence. It includes 8 questions that assess various factors that can affect medication use, such as forgetfulness, busyness and side effects. Scores range from 0 to 8, with lower scores reflecting better adherence.
Time Frame: cross-sectional, 1 hour interview after clinic visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adult Patients With Diabetes and Hypertension: English-speaking, adult patients with diabetes and hypertension were enrolled in the study. There are no study arms.
Arm/Group | Adult Patients With Diabetes and Hypertension
Number analyzed (Participants) | 179
units on a scale
  MeDS tool | 10.9 (2.6)
  Morisky Adherence Measure | 2.5 (1.7)
Statistical Analysis 1: Comparison: Adult Patients With Diabetes and Hypertension; We examined correlations between patient scores on the Measure of Medication Self-Management (MeDS) and the 8-item Morisky Medication Adherence questionnaire; Test type: Superiority or Other; p < .001, Correlation; correlation coefficient = .60 — r= 0.60, p-value<0.001. P values below 0.05 are considered statistically significant in this study

ADVERSE EVENTS:
Time Frame: There is no adverse event reporting. This was a cross sectional study to develop a medication self-management scale.
Groups:
- Adult Patients With Diabetes and Hypertension: There are no study arms. This was a cross-sectional study to develop a medication self-management scale.
Arm/Group | Adult Patients With Diabetes and Hypertension
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less